CLINICAL TRIAL: NCT01824992
Title: a Multi-sites, Randomized, Parallel, Controlled Clinical Study to Evaluated the Efficacy and Safety of Recombinant Human Interferon Alpha-2b Gel (Yallaferon®) in HPV Infection
Brief Title: Recombinant Human Interferon a-2b Gel for HPV Gynecological Infections
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Lee's Pharmaceutical Limited (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: LeesPharm_RHI; China State FDA (Other: China State Food and Drug Administration)
Record Dates: First submitted 2013-03-26; First posted 2013-04-05 (Estimated); Last update posted 2013-04-05 (Estimated); Status verified 2013-04

CONDITIONS: HPV Infection
MeSH Terms: conditions — Papillomavirus Infections

ARMS (2):
- Observation (No Intervention): subject only got observation
- Drug (Experimental): subject were treated with Yallaferon®， the recombinant human interferon α-2b gel
  Interventions: Drug: Yallaferon®

INTERVENTIONS:
Drug: Yallaferon®
  Other Names: Yallaferon®， the recombinant human interferon α-2b gel
  Arms: Drug

SUMMARY:
to assess the efficacy and safety of recombinant human interferon α-2b gel (Yallaferon®) for the treatment of patients with cervical high-risk HPV infections; to analyze the HPV type infections and clinical negative conversion.

285 patients with positive high risk HPV infection were randomized into interferon gel group and control group at ratio of 2:1 (203 patients in treatment group and 82 patients in control group). The patients in treatment group received 1g recombinant human α-2b interferon gel every other day for consecutive 3 courses of treatment, whereas no treatment was conducted in control group.

ELIGIBILITY:
Inclusion Criteria:

1. Age 30 to 65 years of age the sex life of female patients;
2. , liquid-based cytology (TCT) check no intraepithelial lesions and malignant cells;
3. , HPV DNA typing test for high-risk HPV positive (including a single high-risk type positive, and more high-risk type of positive and high-and low-risk hybrid positive).

15 kinds of high-risk types, including HPV16, 18,31,33,35,39,45,51,52,53,56,58,59,66,68

Exclusion Criteria:

* (1) cervical intraepithelial neoplasia (CIN); (2), combined with a severe fungal, trichomonas vaginitis; (3), severe primary diseases associated with cardiovascular, liver, kidney and hematopoietic system; (4), allergies or allergy to the drug known ingredients. (5), within 30 days to accept other clinical trials of drugs or are participating in clinical trials; (6), pregnant and lactating women and to be pregnant women; (7), the researchers do not consider it appropriate clinical trials.

Ages: 30 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 325 (Actual)
Dates: Start 2011-03; Primary Completion 2012-03 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
difference of hr-HPV DNA negative conversion rate | six months
  Primary efficacy endpoint was the difference of hr-HPV DNA negative conversion rate on the 6th month between the two groups.

SECONDARY OUTCOMES:
Secondary efficacy endpoints were the differences of single-type HPV infection, dual infection and multiple infections on the 6th month between the two groups. | six months
  Secondary efficacy endpoints were the differences of single-type HPV infection, dual infection and multiple infections on the 6th month between the two groups.
  Evaluation criteria:
  Negative conversion was defined as all positive hr-HPV DNA at baseline turning negative.
  Non-negative conversion was defined as at least one of the positive hr-HPV DNA at baseline not turning negative.